CLINICAL TRIAL: NCT05793892
Title: A Phase III Clinical Study of the Efficacy and Safety of Lidocaine and Tetracaine Cream (CU-30101) in a Multicenter, Randomized, Double-Blind, Active-Controlled, Paired Design for Facial Laser Aesthetics in Chinese Adults
Brief Title: Efficacy and Safety of Lidocaine and Tetracaine Cream for Facial Laser Aesthetics in Chinese Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CU-30101-304
Record Dates: First submitted 2023-03-09; First posted 2023-03-31 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: test drug：Lidocaine tetracaine cream（CU-30101） control drug：Lidocaine tetracaine cream（Pliaglis®）
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): The order of administration of the test drug in both treatment areas in Arm A is the first, followed by the use of the control drug.
  Interventions: Drug: Lidocaine tetracaine cream
- Arm B (Active Comparator): The order of administration in both treatment areas in Arm B was the use of the control drug first, followed by the investigational drug.
  Interventions: Drug: Lidocaine tetracaine cream

INTERVENTIONS:
Drug: Lidocaine tetracaine cream — The test drug and the control drug will be uniformly spread over the treatment area using a tongue platula to form a thin layer of approximately 1 mm,right then left . The drug remained in the treatment area for 30 minutes (± 2 minutes) .
  Other Names: test drug:CU-30101; control drug:Pliaglis

SUMMARY:
Lattice laser is a new medical cosmetic technology, which is a kind of noninvasive and invasive technology. Compared with traditional laser therapy, lattice laser has a wider range of clinical use, and can be used to treat skin problems such as acne marks, fine wrinkles, skin aging, chloasma, coffee spots, large pores and dullness. Dot-array laser has been widely used in the treatment of skin diseases and skin cosmetics because of its advantages of small trauma, rapid recovery, safety and effectiveness, and fewer complications. The facial skin is rich in nerve fibers and pain receptors are distributed punctuately. Most patients have pain and discomfort to varying degrees during laser treatment. The pain and discomfort associated with laser treatment of the face make anaesthesia an important assistant technique in laser skin cosmetology. At present, the commonly used anesthesia methods to relieve pain include: local cooling anesthesia, topical anesthesia, general anesthesia, gas inhalation anesthesia, intravenous anesthesia, iontophoresis anesthesia, etc. General anesthesia is usually associated with a risk of complications, residual areas of regional nerve block are often sensitive to pain, and acupuncture and drug injection can increase patient discomfort. Therefore, because of its simplicity and convenience of drug administration, topical anesthesia has a positive significance in facial lattice laser cosmetic treatment. The reference product lidocaine tetracaine cream (brand name: Pliaglis ®) has been marketed in the United States and the European Union for many years, and its therapeutic efficacy has been clinically recognized and has a good safety profile.Lidocaine tetracaine cream (R & D code: CU-30101) is manufactured by Cutia Therapeutics (Wuxi) Co., Ltd . A randomized, double-blind, multi-center clinical study is currently proposed to evaluate the efficacy and safety of CU-30101 in facial spot-array laser cosmetology in Chinese subjects with Pliaglis ® as a control.

DETAILED DESCRIPTION:
On the one hand, MTZ can self-repair, stimulate collagen regeneration and improve skin texture; on the other hand, due to the small area of MTZ injury, the surrounding normal skin tissue can be rapidly repaired, reduce the risk of treatment and shorten the recovery time. Lattice laser is a new medical cosmetic technology, which is a kind of noninvasive and invasive technology. Compared with traditional laser therapy, lattice laser has a wider range of clinical use, and can be used to treat skin problems such as acne marks, fine wrinkles, skin aging, chloasma, coffee spots, large pores and dullness. Dot-array laser has been widely used in the treatment of skin diseases and skin cosmetics because of its advantages of small trauma, rapid recovery, safety and effectiveness, and fewer complications. The facial skin is rich in nerve fibers and pain receptors are distributed punctuately. Most patients have pain and discomfort to varying degrees during laser treatment. The pain and discomfort associated with laser treatment of the face make anaesthesia an important assistant technique in laser skin cosmetology. At present, the commonly used anesthesia methods to relieve pain include: local cooling anesthesia, topical anesthesia, general anesthesia, gas inhalation anesthesia, intravenous anesthesia, iontophoresis anesthesia, etc. General anesthesia is usually associated with a risk of complications, residual areas of regional nerve block are often sensitive to pain, and acupuncture and drug injection can increase patient discomfort. Therefore, because of its simplicity and convenience of drug administration, topical anesthesia has a positive significance in facial lattice laser cosmetic treatment. The reference product lidocaine tetracaine cream (brand name: Pliaglis ®) has been marketed in the United States and the European Union for many years, and its therapeutic efficacy has been clinically recognized and has a good safety profile. In accordance with the Chemical Drug Registration Category and Application Dossier Requirements (NMPA 2020 No. 44), lidocaine tetracaine cream (R & D code: CU-30101) manufactured by Corde Biopharmaceuticals (Wuxi) Co., Ltd. is registered as a chemical class 3. A randomized, double-blind, multi-center clinical study is currently proposed to evaluate the efficacy and safety of CU-30101 in facial spot-array laser cosmetology in Chinese subjects with Pliaglis ® as a control.

ELIGIBILITY:
Inclusion Criteria:

* (1) fully informed, fully understand the trial content, process, benefits and possible adverse reactions, and voluntarily participate in the trial, and sign the informed consent;
* 2、Aged 18-65 years old (including the boundary value), gender is not limited;
* (3) Body mass index (BMI) between 18.5-28.0 kg/m2 (including the boundary value);
* (4) plan to perform facial lattice laser cosmetic;
* (5) The subject can communicate well with the investigator and can complete the study in accordance with the provisions of the study.

Exclusion Criteria:

* (1) At screening, the investigator judged that the subject has facial skin damage, peeling, tattoo, scar, atopic dermatitis, urticaria or other skin diseases that may interfere with the study objectives and evaluation;
* (2) sensory disturbance, hyperalgesia, migraine, herpes zoster, trigeminal neuralgia and other head and facial pain affect the efficacy evaluation;
* (3) Those who have used any analgesics within 24 hours before surgery;
* (4) Patients with allergic constitution [to two or with substances (dust, pollen, food, drugs, etc.)], or known to be allergic to lidocaine, tetracaine or other amide or ester local anesthetics and its excipients or p-aminobenzoic acid (PABA);
* (5) Those who are sensitive to systemic effects of lidocaine and tetracaine (such as acute disease, severe liver disease or pseudocholinesterase deficiency);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
the VAS score of immediate pain | after each side lattice laser cosmetic surgery
  The subjects completed the VAS score of immediate pain at the test drug site and the control drug site after each side lattice laser cosmetic surgery;

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Shanghai Ninth People Hospital,Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Beijing Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - West China School of Medicine West China Hospital of sichuan university, Chendu
  - Fujian Medical University Union Hospital, Fuzhou
  - Nanfang Hospital/Guangzhou, Guangzhou
  - Jiangsu Province Hospital, Nanjing
  - Union Hospital, Tongji Medical college huazhong university of science and technology, Wuhan
  - The affiliated hospital of xuzhou medical university, Xuzhou

IPD SHARING:
Plan to Share IPD: No